CLINICAL TRIAL: NCT05922020
Title: The Effect of Hyperoxia on Ventilation During Recovery From General Anesthesia: A Crossover Preliminary Investigation
Brief Title: Hyperoxia on Ventilation During Recovery From General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Anthony Doufas, Professor of Anesthesiology, Perioperative and Pain Medicine, Stanford University
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: IRB-70628
Record Dates: First submitted 2023-06-18; First posted 2023-06-28 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Ventilatory Depression; Postoperative Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — nitrox

STUDY DESIGN:
Intervention Model Description: With the patients' admission to the post-anesthesia care unit and after a 20-minute-long stabilization period, two 40-minute-long treatment sessions will be applied to the study patients. In the first 6 patients Conservative O2 treatment will be applied first, whereas in the rest (patients 7-10) the order of the interventions will be reversed. The order of the interventions will not be revealed to the participants before completing the study. In the Conservative O2 treatment session, O2 supplementation will be titrated to an SpO2 between 90% and 94%, while in the Liberal O2, O2 administration will be titrated to an SpO2 > 96%.
Who Masked: Participant, Outcomes Assessor
Masking Description: 1. Study participants will not be aware of the inspired O2 concentration in their breathing gas mixture. All participants will be breathing through a non-rebreather mask, which will be connected via a Y -piece to both the O2 and air wall outlets.
  2. The investigator who will regulating the O2 inspired concentration-related intervention, will be blinded to the continuous TcPCO2 measurement. In addition, the sleep medicine specialist who will assess the breathing pattern offline and score the number and nature of apnea/hypopnea episodes, will also be blinded to the treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Conservative O2" (Active Comparator): During the first treatment session, which will last for 40 minutes, O2 supplementation will be titrated to an SpO2 between 90% and 94%.
  Interventions: Other: Oxygen gas
- "Liberal O2" (Experimental): During the second treatment session, which will last for 40 minutes, O2 supplementation will be titrated to an SpO2 > 96%.
  Interventions: Other: Oxygen gas

INTERVENTIONS:
Other: Oxygen gas — Administration of Oxygen by inhalation

SUMMARY:
In this preliminary, crossover investigation the investigators will examine the effect of oxygen supplementation on the recovery of breathing in the immediate post-anesthesia period.

DETAILED DESCRIPTION:
In a pilot randomized-controlled trial (NCT04723433) the investigators found that, compared with standard O2 supplementation, hyperoxia enhanced ventilation, as estimated by the fraction of time at a transcutaneous PCO2 (TcPCO2) > 45 mmHg.

More specifically, patients treated with hyperoxia (O2 titrated to: SpO2 > 96%, N=10; Liberal O2) for 90 minutes post-anesthesia, spent 61.2% of the time at TcPCO2 > 45 mmHg, compared with 80.6% of the time in those receiving standard O2 supplementation (O2 titrated to: SpO2 between 90-94%, N=9; Conservative O2 - between-group difference of 19.4% (95% Confidence Intervals: -18.7% to 57.6%), ANCOVA adjusted P = 0.140]. Results were consistent across the 90-min monitoring period. With an observed effect size of 0.73, it was estimated that 30 participants per group are required, to demonstrate this difference with a power of 80% at a two-sided alpha of 5%.

In a follow-up RCT (IRB-63878, NCT05379673) in 18 patients the investigators found that over a 90-minute window, the average percentage of time spent at TcPCO2 > 45mmHg for patients in the Conservative O2 group (N=9) was 57.8% (52 ± 44 minutes), compared with a 45.6% (41 ± 46 minutes) for those in the Liberal O2 group (N=9), (P=0.6134; two-sided two sample t-test). In addition, during the same period, respiratory disturbance index (RDI; events per hour) was higher in the Conservative O2 [median (range): 23.9 (11.0-78.6)], compared with the Liberal O2 group [19.6 (2.8-40.4), Mann-Whitney test, P=0.1615].

Due to the high variability observed in the evaluated respiratory parameters (i.e., TcPCO2 and upper airway obstruction expressed by Respiratory Disturbance Index), the researchers believe that a crossover, rather than a randomized controlled trial, design would improve the power and efficiency of this investigation and also provide an opportunity to characterize better those patients who respond, and separate them from those who do not respond to hyperoxia treatment.

This preliminary investigation will assess how ventilation during recovery from general anesthesia is affected by conservative (Conservative O2: 90% ≤ SpO2 ≤ 94%), compared with liberal (Liberal O2: SpO2 > 96%) O2 supplementation. Using a crossover study design, the investigators aim to: a) assess the breathing pattern and estimate and compare the number of apnea/hypopnea episodes between the two interventions, and b) estimate and compare the cumulative segment of time during which the transcutaneous partial pressure of carbon dioxide (TcPCO2) will exceed 45 mmHg, between the two interventions.

Hypothesis: Conservative O2 will be associated with more unstable and obstructed breathing and less time spent with TcPCO2 > 45 mmHg, compared with Liberal O2 supplementation, during recovery from anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-III
* Body mass index (BMI) less than 35 kg/m2
* Scheduled to undergo robotic-assisted radical laparoscopic nephrectomy.

Exclusion Criteria:

* Patients with a diagnosis of chronic obstructive pulmonary disorder (COPD), severe neurological, cardiopulmonary, psychiatric, or untreated thyroid disorder
* Chronic pain condition that is being treated with opioids
* Patients with a hematocrit lower than 30% at the end of surgery, or those with an excessive blood loss, requiring transfusion of blood products during surgery.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Respiratory disturbance index (RDI) | Forty minutes of monitoring for each treatment arm
  The number of apnea/hypopnea episodes detected using respiratory inductance plethysmography and nasal flow.
Transcutaneous carbon dioxide pressure (TcPCO2) | Forty minutes of monitoring for each treatment arm
  The cumulative segment of time during which the transcutaneous partial pressure of carbon dioxide will exceed an upper limit of 45 mmHg (i.e., TcPCO2 > 45 mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Doufas, MD, PhD, Principal Investigator — Professor, Department of Anesthesiology, Stanford University Medical School
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kutscher S, Finnsson E, Tian L, Panousis P, Chung BI, Doufas AG. The effect of hyperoxia on disordered breathing during recovery from general anesthesia: A single-blinded, crossover, non-randomized -controlled, trial. J Clin Anesth. 2026 Jan;108:112057. doi: 10.1016/j.jclinane.2025.112057. Epub 2025 Oct 31. PMID 41175776